CLINICAL TRIAL: NCT06845319
Title: Anthracycline-Free Neoadjuvant Chemoimmunotherapy for Triple Negative Breast Cancer Patients With Cardiomyopathy or at an Elevated Risk of Cardiotoxicity (NeoCARD): A Response Adapted Single-arm Phase 2 Trial
Brief Title: Anthracycline-Free Neoadjuvant Chemoimmunotherapy for Triple Negative Breast Cancer Patients
Acronym: NeoCARD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104060
Record Dates: First submitted 2025-02-11; First posted 2025-02-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Carboplatin; Paclitaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TNBC + non inflammatory Stage 2 3A/B (Experimental)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin target AUC 5 every 3 weeks for 12-18 weeks OR target AUC 1.5 every week for 12-18 weeks (per investigator's choice).
Drug: Paclitaxel — 80mg/m2 weekly
Drug: Pembrolizumab — 200 mg every 3 weeks for 4 cycles

SUMMARY:
This is a multi-institute, single-arm Phase II study to assess the efficacy of a 12-18-week neoadjuvant carboplatin, paclitaxel, and pembrolizumab (CPP) regimen in a response-adaptive manner for triple-negative breast cancer (TNBC) patients who are ineligible for anthracycline-based therapy due to underlying cardiac conditions.

DETAILED DESCRIPTION:
Clinical trial participation among patients with cardiac co-morbidities is limited, creating challenges for oncologists managing aggressive cancers like Triple Negative Breast Cancer (TNBC) in this demographic. At MUSC and its rural sites, a significant patient population faces such complexities, particularly African Americans (AA) who are predisposed to anthracycline-induced cardiotoxicity. Hence, proposing a dedicated study targeting patients with cardiomyopathy or at high cardiotoxicity risk, utilizing a non-anthracycline regimen, is essential.

Rationale for Using Taxol, and Carboplatin with Immunotherapy:

It is estimated that around 60% of TNBC patients exhibit a "BRCAness" phenotype, which mirrors the clinical characteristics of tumors with BRCA mutations. Consequently, the use of DNA-damaging agents, like platinum-based therapies, has gained prominence as a viable treatment option for these patients. Several studies have demonstrated that adding carboplatin to neoadjuvant chemotherapy regimens improves the pathological complete response rates in TNBC patients. While some trials have also shown improvements in disease-free survival, others have not observed this benefit. Notably, a recent study from India highlighted an overall survival advantage, specifically in TNBC patients under the age of 50, when carboplatin was included in their treatment.

Taxanes are well-established in improving pathologic complete response (pCR) rates, which are strongly correlated with better long-term outcomes in TNBC. Emerging evidence suggests that taxanes may also enhance antitumor immune responses, making them an excellent partner for immune checkpoint inhibitors in TNBC.

Studies have demonstrated that taxanes increase the proliferation of CD8-positive T cells and enhance the recruitment of tumor-infiltrating lymphocytes (TILs), both of which contribute to improved tumor cell apoptotic responses. Furthermore, paclitaxel has been shown to directly influence dendritic cell activity. It promotes the upregulation of cation-independent mannose-6-phosphate receptors on the surface of tumor cells, thereby enhancing the efficacy of granzyme B-mediated cytotoxic killing of tumor cells.

This dual mechanism-direct tumor cytotoxicity and immune modulation-highlights the versatility and importance of taxanes in combination therapies for TNBC, particularly in regimens incorporating immunotherapy.

Platinums have also been shown to modulate the immune system and cause immunogenic mediated cell death whereby they can increase major histocompatibility complex (MHC) class I expression on cancer cells thus promoting T-cell activation. Although platinums on their own could induce an immune response, a combination with taxanes like paclitaxel has been shown to augment this response as evidenced by decreasing T regulatory cells and increasing the proportions of T-helper cells and natural killer cells. In a mouse study looking at combining cisplatin with paclitaxel and immunotherapy, it was found that chemotherapy enhanced immune-mediated cancer cell death by decreasing intratumoral T regulatory cells and increasing the recruitment of cytokine-induced killer cells.

Rationale for Weekly Taxol Over Taxotere:

In the ECOG 1199 trial, two taxanes, paclitaxel, and docetaxel, were compared in two regimens, weekly or every 3 weeks, alongside Adriamycin Cytoxan. Overall survival favored weekly paclitaxel over every 3-week paclitaxel (OR 1.32, P=0.01). After 12.1 years, both weekly paclitaxel and every 3-week docetaxel remained linked to improved disease-free survival (DFS) and slightly better overall survival (OS) compared to every 3-week paclitaxel. Among 1025 TNBC patients, weekly paclitaxel emerged as the most effective taxane. Ten-year progression-free survival (PFS) with weekly paclitaxel increased to 69% from 62% with every 3-week docetaxel (P=0.032), while ten-year OS rose to 75% from 69% (P=0.094).

In terms of chemotherapy-related toxicities, every 3-week docetaxel was associated with higher levels of grade 4 toxicities than weekly paclitaxel 50% versus 4% respectively and most of the side effects are related to grade 4 neutropenia (46% vs 2%), febrile neutropenia (16% vs 1%), grade 3-4 stomatitis, fatigue, and myalgias. Conversely, the paclitaxel group had a higher level of grade 3 or 4 neuropathy of around 8% versus 4%. Unique to docetaxel, patients can also experience fluid retention syndrome often requiring prophylaxis with corticosteroids. This can manifest as peripheral edema, pleural effusions, ascites, or generalized weight gain. The condition is dose-dependent and typically more pronounced in patients receiving higher cumulative doses of docetaxel.

Rationale for a 12-Week Regimen:

The effectiveness of regimens featuring weekly taxanes with carboplatin is highlighted in studies like the WSG-ADAPT TN study and the phase 2 study by Loi et al, which show better tolerance among patients with underlying health conditions. A 12-week platinum/taxane/pembrolizumab protocol may achieve pathological complete response (pCR) in chemo-sensitive patients without the need for prolonged chemotherapy. However, individuals with poor response rates may require extended therapy. Early identification of responders through radiographic methods could enable de-escalation strategies, potentially reducing long-term toxicities such as neuropathy that significantly impact quality of life.

Rationale for Response Adaptive Study Design:

MRI stands out as the most accurate imaging modality for assessing pCR in TNBC patients, with reported accuracy rates exceeding 86%. Therefore, MRI is endorsed as the optimal tool for assessing response by the American College of Radiology (ACR) and the Society of Breast Imaging (SBI)

As assessed by MRI, tumor response to neoadjuvant therapy has been associated with long-term outcomes, such as recurrence-free survival and overall survival. Therefore, adaptive MRI response therapy provides valuable prognostic information to guide post-surgical management and long-term follow-up strategies.

Overall, MRI response adaptive neoadjuvant therapy in breast cancer provides early detection of changes in tumor size and morphology, facilitating prompt assessment of treatment response. Additionally, MRI findings, including alterations in tumor enhancement patterns, can predict pathologic response to therapy, informing decisions about achieving a complete response. These MRI results also guide tailored treatment planning, determining the necessity of additional therapy and suitability for breast-conserving surgery versus mastectomy.

Rationale for the Study Population:

At MUSC and the National Cancer Institute Community Oncology Research Program for Minority-Underserved (NCORP-MU) sites, a substantial proportion of AA patients with multiple cardiac risk factors cannot receive anthracycline-based treatment, revealing a healthcare gap necessitating targeted research. Patients with cardiac comorbidities are frequently excluded from Phase 3 clinical trials, resulting in a significant gap in evidence-based treatment options for this population. Consequently, in current practice, providers often rely on non-anthracycline-based regimens for patients with underlying cardiomyopathy. However, the selection of these regimens is highly variable, with no standardized approach, leading to inconsistent practices across institutions. Moreover, the efficacy, response rates, and tolerability of these regimens remain largely unvalidated, as they have not been systematically studied in formal clinical trials. This lack of high-level evidence highlights the urgent need for dedicated research to establish uniform and effective treatment strategies for this vulnerable group. Clinical calculators have been developed to assess the risk of congestive heart failure in these patients exposed to anthracyclines providing valuable guidance for risk stratification. One such tool, developed by Ezaz et al., utilizes clinical factors to predict CHF risk in cancer patients undergoing treatment. According to this risk prediction model, patients classified as medium risk and high risk have 3-year CHF rates of 26% and 39.5%, respectively, when treated with anthracyclines or trastuzumab. These findings highlight the importance of individualized risk assessment in optimizing treatment strategies for vulnerable populations. This calculator's effectiveness was further confirmed by Milks et al. in a separate cohort of patients undergoing treatment with anthracyclines, with or without trastuzumab.

Hence, investigators propose a pragmatic Phase 2 single-arm study focusing on individuals with T1c, N0, Stage 2, and 3A/B TNBC either afflicted with cardiomyopathy or at elevated risk of cardiotoxicity. These participants will undergo a response-adaptive NAC regimen lasting 12-18 weeks, comprising carboplatin, weekly paclitaxel, and pembrolizumab (CPP).

Rationale for Including Low ER Patients:

The American Society of Clinical Oncology and the College of American Pathologists (ASCO/CAP) defined ER-positive breast cancer as ER ≥ 1% of stained tumor nuclei by IHC. ER expression between 1-10% is classified as ER-low. Despite the above designation, breast tumors that are ER-low behave more like triple-negative tumors. A study at Dana Farber Brigham Cancer Center looked at patients with ER low and correlated it with PAM 50 and Oncotype DX breast recurrence score (RS) when evaluated. Among the ER-low and HER2-negative tumors, 82.6% were basal-like in histology, and 67% had RS ≥ 26; thereby supporting the notion that ER-low tumors tend to be similar to triple-negative tumors in biology. Sharma et al. evaluated 516 patients that represented stage I-3 patients with HER2 negative breast cancer and ER/PR ≤ 10%, and TNBC patients with TNBC defined as ER/PR<1%. RFS and OS between both groups were not significantly different: 3-year RFS 82.5% versus 82.4% and 3-year-OS 88% versus 83.4% respectively.

A retrospective study at MD Anderson Cancer Center that included over 9000 patients, and with a median follow-up of 5.1 years, reported that patients with ER 1-9% had worse survival rates than those with ER ≥ 10% when survival outcomes were not significantly different between ER low and ER-negative tumors.

Despite all of that, patients with ER-low disease tend to be excluded from triple-negative breast cancer studies. Because of their close biology and clinical outcomes, investigators elected to include patients with ER low disease in a triple-negative breast study.

ELIGIBILITY:
Inclusion Criteria:

1. Measurable or evaluable tumor in the breast larger than 1cm with or without axillary involvement.
2. Ability to be followed by a cardiologist and/or primary care physician (PCP) for medication optimization of cardiac co-morbidities.
3. Medically fit to undergo curative surgery as per the standard of care.
4. Ability and willingness to comply with all study procedures.
5. Ability and willingness to sign and date a written informed consent.
6. Female or Male.
7. Age 18 and above.
8. Histologically confirmed TNBC Stage II or Stage IIIA/B.

   1. The invasive tumor must be hormone receptor-negative or low, defined as both estrogen receptor (ER) and or progesterone receptor (PR) staining present in <10% of invasive cancer cells by IHC.
   2. HER2 negativity will be based on current ASCO-CAP guidelines for HER2 testing.
9. In patients with multifocal disease, all the tumors should be HER2-negative.
10. No previous chemotherapy, immunotherapy, radiation therapy, or surgery for this breast cancer.
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
12. Have adequate organ function at the time of screening visit as defined below:

    a. Hematological: i. Absolute neutrophil count ≥ 1,500/uL ii. Platelets ≥ 100,000/uL iii. Leukocytes ≥ 3,000/uL iv. Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (criteria must be met without erythropoietin dependency and without packed red blood cell transfusion within last 2 weeks).

    b. Renal: i. Creatinine ≤ 1.5 mg/dL and/or creatinine clearance ≥ 50 mL/min.

1. Patients with a creatinine clearance (CrCl) between 30 and 50 mL/min may be eligible for the study at the discretion of the Principal Investigator. Given that paclitaxel is primarily metabolized by the liver and not significantly affected by renal function, and that carboplatin dosing can be safely adjusted based on CrCl, enrollment of these patients is permissible following individual assessment and approval.

c. Hepatic: i. Total bilirubin ≤ 1.5x IULN, OR direct bilirubin ≤ IULN for participants with total bilirubin levels > 1.5x IULN. Participants with a history of Gilbert's disease must have total bilirubin ≤ 5x IULN. ii. AST(SGOT) and ALT(SPGT) ≤ 2.5x IULN.

d. Coagulation: i. International normalized ratio (INR) of coagulation OR prothrombin time (PT) OR activated partial thromboplastin time (aPTT) ≤ 1.5x IULN unless the patient is receiving anticoagulant therapy. If the patient is receiving anticoagulant therapy, PT or PTT is within the therapeutic range of the intended use of anticoagulants. e. Serum albumin ≥ 3.0 g/dL. 13. Patients with clinically and/or radiologically abnormal axillary lymph nodes should have pathological confirmation with image-guided biopsy/fine needle aspiration. 14. Patients should have staging scans to exclude the possibility of metastatic disease when axillary imaging shows two or more abnormal lymph nodes, if there are clinical signs concerning for metastatic disease or at the treating physician's discretion. Patients with bilateral breast cancer are eligible if they meet other eligibility criteria and both tumors are HER2 negative.

15. Baseline neuropathy grade ≤2. 16. A WOCBP must be willing and able to use highly effective contraception from the time of informed consent throughout the study period and at least six months after the last dose of trial treatment.

17. Patient is ineligible for anthracycline treatment, as of at least one of the following of A, B, C, or D: A. Individuals identified as being at high risk for cardiotoxicity from anthracycline treatment.

1. Preexisting cardiomyopathy with Ejection Fraction (EF) between 25-49%.
2. Severe valvular disease on echocardiogram.
3. Previous exposure to Anthracyclines.
4. Previous exposure to high dose chest wall radiation >30Gy.
5. Participants who have experienced myocardial infarction, unstable angina pectoris, an arterial thrombotic event, or stroke, within the last 12 months but not less than 3 months ago. B. Medium and High Risk for Congestive Heart Failure (CHF) at 3 years as defined by the Cardiotoxicity prediction tool from Ezaz et al C. Patients declining anthracycline therapy after thorough discussion regarding its significant role in treating TNBC. D. Patients who are deemed ineligible for anthracycline due to underlying medical conditions, as determined by the primary oncologist and confirmed by the study PI.

18. Breast and axillary imaging (including ultrasound and MRI) within 42 days (6 weeks) prior to registration.

Exclusion Criteria:

1. Subject is planning to participate, currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
2. Current diagnosis of metastatic or inflammatory breast cancer.
3. Patients deemed unfit to undergo curative surgery according to the standard of care.
4. Patients who have concomitant and/or previous malignancies within the last 5 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., ductal carcinoma in situ (DCIS), carcinoma in situ of the cervix) that have undergone potential curative therapy are NOT excluded.
5. History of hypersensitivity to compounds that are similar to carboplatin and paclitaxel
6. Has received major surgery and has not recovered adequately from the toxicity and/or complications before starting study treatment.
7. Subject has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza or COVID vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy (7-day clearance period for immunosuppressant therapy prior to starting study treatment, if applicable).
9. Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e., with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
10. Has a history of solid organ transplant.
11. Has a history of non-infectious pneumonitis that required high-dose steroids and/or has current pneumonitis.
12. Has an active bacterial infection requiring systemic therapy.
13. History of Human Immunodeficiency Virus (HIV).
14. History of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as detectable HCV RNA) infection.
15. Known psychiatric or substance abuse disorders that would interfere with the requirements of the trial.
16. Pregnant or breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment.
17. Subject is a WOCBP who has had a positive urine pregnancy test within 24 hours prior to initiation of study treatment. Females will be determined to be not of child-bearing potential with a history of hysterectomy or with postmenopausal status of >12 months.
18. Uncontrolled hypertension (systolic BP > 180 bpm or diastolic BP > 100 bpm), or uncontrolled or symptomatic arrhythmia at the time of screening visit.
19. At time of screening visit, EF less than 25%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2027-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
pCR Rate in TNBC patients | 18 weeks
  To determine the pCR rate in TNBC patients treated with the 12-18 weeks CPP regimen

SECONDARY OUTCOMES:
Radiological Response | 12 weeks
  To evaluate radiologic response rate (RRR) at 12-week MRI defined by complete response and partial response.
Minimal Residual Disease Rate | 18 Weeks
  To evaluate the minimal residual disease (MRD) rate (residual cancer burden score of 0+1) with the neoadjuvant CPP regimen
Event Free Survival | 3 years
  To determine 3-year event-free survival (EFS) with a neoadjuvant CPP regimen
Overall Survival | 5 years
  To determine 3 and 5-year overall survival (OS) with a neoadjuvant CPP regimen
Quality of life of patients with cardiac conditions undergoing the CPP regimen. | 5 years
  Quality of life (QOL) will be evaluated using PROMIS-29 Profile v2.1 at baseline, at the conclusion of NAC and again at 12 months postNAC.
To evaluate the toxicity of neoadjuvant CPP regimen in TNBC patients with underlying cardiac conditions | 5 years
  Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.03. Start of study treatment (cycle 1 day 1) until 30 days after last dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Abi Siva, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States